CLINICAL TRIAL: NCT03924089
Title: Effect of an Oral Nutritional Supplement on Nutritional and Functional Status, Biological Markers (Inflammation and Oxidative Stress, Intestinal Microbiota, Circulating microRNA and Its Target Genes) in Malnourished Hemodialysis Patients.
Brief Title: Oral Nutritional Supplement on Nutritional and Functional Status, and Biomarkers in Malnourished Hemodialysis Patients.
Acronym: RENACARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI18/01041
Record Dates: First submitted 2019-04-08; First posted 2019-04-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-02

CONDITIONS: Malnutrition; End Stage Renal Disease
MeSH Terms: conditions — Malnutrition; Kidney Failure, Chronic | interventions — Dietary Supplements; Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, parallel-group trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open to the intake of ONS or diet, but double-blind to the intake of probiotics
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral nutritional supplement with probiotics (Experimental): Oral nutritional supplement specifically developed for undernourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants, carnitine), with probiotics.
  Physical activity recommendations.
  Interventions: Dietary Supplement: Oral nutritional supplement with probiotics
- Oral nutritional supplement without probiotics (Experimental): Oral nutritional supplement specifically developed for undernourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants, carnitine), without probiotics.
  Physical activity recommendations.
  Interventions: Dietary Supplement: Oral nutritional supplement without probiotics
- Individualized dietary recommendations (Active Comparator): Individualized dietary recommendations. Physical activity recommendations.
  Interventions: Other: Dietary recommendations

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement with probiotics — Oral nutritional supplement specifically developed for undernourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants and carnitine), with probiotics.
  Other Names: Physical activity recommendations.
  Arms: Oral nutritional supplement with probiotics
Dietary Supplement: Oral nutritional supplement without probiotics — Oral nutritional supplement specifically developed for undernourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants and carnitine), without probiotics.
  Other Names: Physical activity recommendations.
  Arms: Oral nutritional supplement without probiotics
Other: Dietary recommendations — Dietary recommendations
  Other Names: Physical activity recommendations.
  Arms: Individualized dietary recommendations

SUMMARY:
Malnutrition in hemodialysis patients is frequent and it is associated with a reduction in muscular mass, strength, functional capacity and quality of life, with an increment in inflammatory and oxidative markers, and with a dysregulation of circulating miRNAs and its target genes.

Animal and human studies have reported that some dietary components (macronutrients, micronutrients and other bioactive substances) might restore these altered features.

Thus, we hypothesized that the intake of an oral nutritional supplement (ONS) specifically developed for malnourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants, carnitine, and with or without probiotics) vs. individualized diet recommendations might:

* Improve nutritional status (visceral proteins, muscular mass), functional capacity and quality of life.
* Reduce inflammatory and oxidative markers, and modulate the circulating levels of some miRNAs and the expression of its target genes on cells. miRNAs may be useful biomarkers to check the response to a nutritional intervention in malnourished hemodialysis patients.

The present study is a randomized, multicenter, parallel-group trial with 3 groups, open to the intake of ONS or individualized diet recommendations, but double-blind to the intake of probiotics. Inclusion criteria comprised adult subjects (>18 y/o) undergoing hemodialysis more than 6 months previous at inclusion and at least one of these caloric malnutrition criteria: a) involuntary weight loss >5% in 3 months or >10% in 6 months; b) serum albumin < 3.5 g/dl or prealbumin <28 mg/dl; c) body mass index (BMI) < 23 kg/m2; d) muscular mass loss >5% in 3 months or >10% in 6 months.

The study duration is 6 months, and comprises 4 visits (screening, basal, 3 months and 6 months). A nutritional examination that included anthropometric measurements, handgrip strength measured by a hand dynamometer, body composition assessed by bioelectrical impedance analysis (BIA) and a 5 days dietary record; quality of life evaluation by the "12-item short form health survey"; the presence of symptoms of depression and anxiety (Hospital Anxiety and Depression Scale); assessment of functional status by the "Barthel" test, the "Short Physical Performance Battery" and the "International Physical Activity Questionnaire"; and blood and stool samples will be obtained for each participant in each study visit (except screening visit).

DETAILED DESCRIPTION:
Hypothesis:

The intake of an oral nutritional supplement (ONS) specifically developed for malnourished hemodialysis patients enriched with functional nutrients (extra virgin olive oil, omega 3 fatty acids, whey protein, antioxidants, carnitine, and with or without probiotics) vs. individualized diet recommendations might:

* Improve nutritional status (visceral proteins, muscular mass), functional capacity and quality of life.
* Reduce inflammatory and oxidative markers, and modulate the circulating levels of some miRNAs and the expression of its target genes on cells. miRNAs may be useful biomarkers to check the response to a nutritional intervention in undernourished hemodialysis patients.

Aims:

To evaluate:

* The clinical response after the nutritional intervention:

  1. Nutritional status: anthropometric measurements, handgrip strength measured by a jamar hand dynamometer, body composition assessed by bioelectrical impedance analysis (BIA), and a 5 days dietary record.
  2. Functional status assessed by the "Barthel" test, the "Short Physical Performance Battery" and the "International Physical Activity Questionnaire".
  3. Quality of life assessed by the "12-item short form health survey", and the presence of symptoms of depression and anxiety by the "Hospital Anxiety and Depression Scale".
* The physiological response after the nutritional intervention:

  1. Inflammatory markers.
  2. Oxidative markers.
  3. Gut microbiota.
  4. Circulating miRNAs and the expression of its target genes on cells.

Study design:

* Randomized, multicenter, parallel-group trial with 3 groups, open to the intake of ONS or diet, but double-blind to the intake of probiotics.
* Study centers:

  1. Hospital Regional Universitario de Málaga (Spain).
  2. Hospital San Cecilio. Granada (Spain).
  3. Hospital Rey Juan Carlos. Móstoles, Madrid (Spain).
* One-hundred and twenty patients will be included. Eligible subjects will be invited to participate, and written informed consent will be obtained before the inclusion. Participants will be randomly assigned to one of these three groups:

  1. ONS with probiotics. Dietary and physical activity recommendations.
  2. ONS without probiotics. Dietary and physical activity recommendations.
  3. Dietary and physical activity recommendations.
* The study duration is 6 months, and comprises 4 visits (screening, basal, 3 months and 6 months). Recruitment period: 12 months.
* Inclusion criteria: adult subjects (>18 y/o) undergoing hemodialysis more than 6 months previous at inclusion and at least one of these caloric malnutrition criteria: a) involuntary weight loss >5% in 3 months or >10% in 6 months; b) serum albumin < 3.5 g/dl or prealbumin <28 mg/dl; c) body mass index (BMI) < 23 kg/m2; d) muscular mass loss >5% in 3 months or >10% in 6 months.
* A nutritional examination that included anthropometric measurements, handgrip strength measured by a jamar hand dynamometer, body composition assessed by bioelectrical impedance analysis (BIA) and a 5 days dietary record; quality of life evaluation by the "12-item short form health survey"; the presence of symptoms of depression and anxiety (Hospital Anxiety and Depression Scale); assessment of functional status by the "Barthel" test, the "Short Physical Performance Battery" and the "International Physical Activity Questionnaire"; and blood and stool samples will be obtained for each participant in each study visit (except screening visit).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (>18 y/o) undergoing hemodialysis more than 6 months previous at inclusion.
* At least one of these caloric malnutrition criteria: a) involuntary weight loss >5% in 3 months or >10% in 6 months; b) serum albumin < 3.5 g/dl or prealbumin <28 mg/dl; c) body mass index (BMI) < 23 kg/m2; d) muscular mass loss >5% in 3 months or >10% in 6 months.
* Standard hemodialysis therapy (3 days/week, 240 min, high permeability dialyzer, blood flow >250 ml/min and dialysate flow 500 ml/min) or on-line hemodialysis therapy that was not modified in the last 3 months previous to the inclusion.
* Written informed consent obtained.

Exclusion Criteria:

* Type 1 diabetes mellitus or type 2 diabetes mellitus with HbA1c>9%.
* Unstable dry weight.
* Limb amputation.
* Significant edema.
* Active malignancy.
* Hospital admissions in the last 3 months.
* Acute gastrointestinal disease in the 2 weeks before the inclusion.
* Gastrectomy, gastroparesis or abnormal gastric emptying.
* Acute heart failure grade IV.
* Severe hepatic insufficiency (men gamma glutamyl transferase -GGT- >150 U/l, women >120 U/l).
* Alcohol or other drugs abuse.
* Participants enrolled in other research study at inclusion.
* Pregnant women.
* No informed consent obtained.
* Patients who received any oral nutritional supplement (specific for hemodialysis patients or not) in the 4 weeks before the inclusion.
* Patients receiving enteral tube feeding.
* Galactosemia, fructosemia, or requirement of a no fiber diet.
* Allergy or hypersensitivity to any ingredient of the oral nutritional supplement.
* Ongoing treatment with glucocorticoids.
* Patients who received any oral fatty acids omega-3 supplement in the 4 weeks before the inclusion.
* Patients who received intradialytic parenteral nutrition in the 3 months before the inclusion.
* Patients who received any probiotics or prebiotics (not as part of the diet) in the 3 months before the inclusion.
* Anemia (Hemoglobin < 10 g/dl) or Epoetin resistance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline and 6 months
  Weight in kg
Change in fat free body mass | Baseline and 6 months
  Fat free body mass in kg assessed by bioelectrical impedance analysis
Change in serum albumin concentration | Baseline and 6 months
  Serum albumin in g/dl
Change in serum prealbumin concentration | Baseline and 6 months
  Serum prealbumin in mg/dl

SECONDARY OUTCOMES:
Change in handgrip strength | Baseline and 6 months
  Handgrip strength in kg, measured by the jamar hydraulic hand dynamometer.
Change in the score of the "Barthel" test. | Baseline and 6 months
  The Barthel is a 10-item ordinal scale that measures functional independence in the domains of personal care and mobility. Specifically, it measures self-care, sphincter management, transfers and locomotion. The score ranges between 0 and 100 points. Scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, 91-99 indicates "slight" dependency, and 100 indicates independency.
Change in the score of the Hospital Anxiety and Depression Scale (HADS). | Baseline and 6 months
  Symptoms of depression and anxiety assessed by the Hospital Anxiety and Depression Scale (HADS). This questionnaire comprises two sub-scales, each one range from 0 to 21 points; one assesses the symptoms of depression, and the other one the symptoms of anxiety. At each sub-scale, a score below 7 is considered normal range, between 8 and 10 means probable presence of depression or anxiety respectively, and more than 11 suggests the presence of depression or anxiety respectively.
Changes in plasma levels of high sensitivity C reactive protein (hs-CRP) | Baseline and 6 months
  Plasma levels of high sensitivity C reactive protein (hs-CRP) in mg/dl
Changes in plasma levels of 8-iso-prostaglandina F2 α (8-iso-PGF2-α) | Baseline and 6 months
  Plasma levels of 8-iso-prostaglandina F2 α (8-iso-PGF2-α) in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira, MD, PhD, Principal Investigator — Instituto de Investigación biomédica de Málaga
Locations (3):
- Spain (3):
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital San Cecilio, Granada
  - Hospital Regional Universitario de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No
The data will be published when the trial will be finished.

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Hevilla F, Padial M, Blanca M, Barril G, Jimenez-Salcedo T, Ramirez-Ortiz M, Nogueira A, Gentile A, Garcia-Escobar E, Romero-Zerbo SY, Olveira G. Effect on nutritional status and biomarkers of inflammation and oxidation of an oral nutritional supplement (with or without probiotics) in malnourished hemodialysis patients. A multicenter randomized clinical trial "Renacare Trial". Front Nutr. 2023 Feb 3;10:1107869. doi: 10.3389/fnut.2023.1107869. eCollection 2023. PMID 36819685
- [Derived] Nishioka N, Luo Y, Taniguchi T, Ohnishi T, Kimachi M, Ng RC, Watanabe N. Carnitine supplements for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013601. doi: 10.1002/14651858.CD013601.pub2. PMID 36472884